CLINICAL TRIAL: NCT00949403
Title: An Interdisciplinary Approach to the Study of Non-alcoholic Fatty Liver Disease
Brief Title: Liver Positron Emission Tomography (PET) Study of Non Alcoholic Fatty Liver Disease
Acronym: Liver
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0621
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Fatty Liver
Keywords: Non-Alcoholic Fatty Liver disease
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Obese Females (pre-bariatric surgery) (Experimental): Twenty obese females (18-45 years of age, BMI > or equal to 45) who are scheduled to undergo bariatric surgery at Barnes-Jewish Hospital will be screened for enrollment over 2 years. They will be imaged with PET/CT and radiopharmaceuticals C-11 Acetate and C-11 Palmitate will be injected.
  Interventions: Drug: Radio pharmaceuticals C-11 Acetate, and C-11 Palmitate

INTERVENTIONS:
Drug: Radio pharmaceuticals C-11 Acetate, and C-11 Palmitate — injection of C-11 Palmitate and C-11 Acetate during PET/CT to determine Liver metabolism

SUMMARY:
The purpose of this study is to evaluate how the liver receives and uses fats for energy. This will help the investigators further understand the physical and chemical processes responsible for Non-Alcoholic Fatty Liver Disease (NAFLD) in overweight females with or without NAFLD who are scheduled to undergo gastric bypass surgery.

DETAILED DESCRIPTION:
This study involves a multidisciplinary approach that will address the metabolic mechanisms responsible for Non-alcoholic Fatty Liver Disease (NAFLD) in humans. Nonalcoholic fatty liver disease (NAFLD) has become an important public health problem in many industrialized countries because of its high prevalence, potential progression to severe liver disease, and association with cardiometabolic abnormalities, including diabetes, the metabolic syndrome, dilated cardiomyopathy, and coronary heart disease. Although obesity is an important risk factor for NAFLD many obese persons have minimal or no steatosis. The mechanism responsible for the pathogenesis of steatosis is not known, but must involve one or more of the following:

1. Increased hepatic fatty acid (FA) delivery
2. Decreased hepatic FA oxidation
3. Increased de novo lipogenesis (DNL)
4. Inadequate hepatic triglyceride secretion

We hypothesize that alterations in all of these metabolic processes are involved in the pathogenesis of NAFLD. However, a comprehensive evaluation of these factors in individual cohorts of subjects has never been performed, and the ability to measure hepatic FA oxidation in vivo in human subjects has not been available.

The following Specific Aims will be evaluated in obese women with and without NAFLD, who are scheduled for bariatric surgery:

1. Determine hepatic FA uptake and oxidation by using novel PET techniques in combination with measurements of DNL using stable isotope tracers and by assessing liver tissue FA oxidative capacity by evaluating gene expression of FA oxidative enzymes and mitochondrial content.
2. Determine hepatic fatty acid delivery by using stable isotope tracers to assess the rate of free FA (FFA) release into plasma and cellular biology methods to determine the expression and protein content of the major tissue FA transporter (CD36).
3. Determine hepatic very-low-density lipoprotein TG (VLDL-TG) secretion rate by using stable isotope tracers.
4. Determine liver histology and factors involved in inflammation and fibrosis by using routine staining and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Obese females with a BMI of greater then or equal to 45.
* Age range between 18-45 years.
* Patients undergoing bariatric surgery at Barnes-Jewish Hospital-St.Louis,MO.

Exclusion Criteria:

* Any prior history or evidence of liver disease other than Non-Alcoholic Fatty liver Disease, severe hypertriglyceridemia and diabetes mellitis.
* Consumed greater then or equal to 20 grams of alcohol per day.
* Taking medications that are known to cause hepatic steatosis & liver damage.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Gropler, MD, Principal Investigator — PI
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Obese Females (Pre-bariatric Surgery): Twenty obese females (18-45 years of age, BMI > or equal to 45) who are scheduled to undergo bariatric surgery at Barnes-Jewish Hospital will be screened for enrollment over 2 years.
Period: Overall Study
Arm/Group | Obese Females (Pre-bariatric Surgery)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution, all efforts to locate the data have been exhausted and therefore no results are available to be reported
Arm/Group | Obese Females (Pre-bariatric Surgery)
Number analyzed (Participants) | 0
Age, Categorical
Age, Categorical
Age, Categorical
Age, Categorical
Age, Categorical
Age, Categorical
Sex/Gender, Customized
Sex/Gender, Customized
Sex: Female, Male
Sex: Female, Male
Obese Females
fatty acid in non-alcoholic Fatty Liver Disease

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fatty Acid Oxidation
Description: Liver fatty acid oxidation as determined by 1-11C-palmitate PET imaging.
Time Frame: 3 hours
Population: as for baseline characteristics
Arm/Group | Obese Females (Pre-bariatric Surgery)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1-2 days
Arm/Group | Obese Females (Pre-bariatric Surgery)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
there were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes